CLINICAL TRIAL: NCT02704533
Title: Sequential Optimization of Dose and Schedule of PfSPZ Vaccine, Verified by Randomized, Controlled, Double-blind Immunization and Controlled Human Malaria Infection in Malaria-naïve, Healthy Adult Volunteers in Germany
Brief Title: Sequential Optimization of Dose and Schedule of PfSPZ Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanaria Inc. (Industry)
Collaborators: Institute of Tropical Medicine, University of Tuebingen (Other); German Federal Ministry of Education and Research (Other Government); German Center for Infection Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MAVACHE; 2015-005123-11 (EudraCT Number)
Record Dates: First submitted 2016-03-01; First posted 2016-03-10 (Estimated); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Malaria
Keywords: Plasmodium falciparum; PfSPZ Vaccine; PfSPZ Challenge (NF54); PfSPZ Challenge (7G8); CHMI
MeSH Terms: conditions — Malaria; Malaria, Falciparum | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (13):
- Optimization Phase - Group A (Experimental): n=6; three times 9x10^5 PfSPZ Vaccine on Days 0, 7 and 28 by DVI. Group A will undergo homologous CHMI with 3,200 PfSPZ Challenge (NF54), 3 weeks after the last dose of vaccine.
  If >75% efficacious, the treatment will be simplified to two times 1.35x10^6 PfSPZ Vaccine on Days 0 and 7 (Group B1).
  If <75% efficacious, the treatment will be increased to three times 1.35x10^6 PfSPZ Vaccine on Days 0, 7 and 28 (Group B2)
  Interventions: Biological: PfSPZ Vaccine; Biological: PfSPZ Challenge (NF54)
- Optimization Phase - Group B1 (Experimental): n=6; two times 1.35x10^6 PfSPZ Vaccine on Days 0 and 7 by DVI. Group B1 will undergo homologous CHMI with 3,200 PfSPZ Challenge (NF54), 3 weeks after the last dose of vaccine.
  If >75% efficacious, the treatment will be simplified to one injection 2.7x10^6 PfSPZ Vaccine (Group C1).
  If <75% efficacious, the treatment will be increased to two times 2.7x10^6 PfSPZ Vaccine on Days 0 and 7 (Group C2).
  Interventions: Biological: PfSPZ Vaccine; Biological: PfSPZ Challenge (NF54)
- Optimization Phase - Group B2 (Experimental): n=6; three times 1.35x10^6 PfSPZ Vaccine on Days 0, 7 and 28 by DVI. Group B2 will undergo homologous CHMI with 3,200 PfSPZ Challenge (NF54), 3 weeks after the last dose of vaccine.
  If >75% efficacious, the treatment will be simplified to two times 2.7x10^6 PfSPZ Vaccine on Days 0 and 7 (Group C2).
  If <75% efficacious, the treatment will be increased to three times 2.7x10^6 PfSPZ Vaccine on Days 0, 7 and 28 (Group C3).
  Interventions: Biological: PfSPZ Vaccine; Biological: PfSPZ Challenge (NF54)
- Optimization Phase - Group C1 (Experimental): n=6; one time 2.7x10^6 PfSPZ Vaccine by DVI. Group C1 will undergo homologous CHMI with 3,200 PfSPZ Challenge (NF54), 3 weeks after vaccination.
  If Group C1 gets vaccinated, study will proceed to verification phase after completion.
  Interventions: Biological: PfSPZ Vaccine; Biological: PfSPZ Challenge (NF54)
- Optimization Phase - Group C2 (Experimental): n=6; two times 2.7x10^6 PfSPZ Vaccine by DVI. Group C2 will undergo homologous CHMI with 3,200 PfSPZ Challenge (NF54), 3 weeks after vaccination.
  If Group C2 gets vaccinated, study will proceed to verification phase after completion.
  Interventions: Biological: PfSPZ Vaccine; Biological: PfSPZ Challenge (NF54)
- Optimization Phase - Group C3 (Experimental): n=6; three times 2.7x10^6 PfSPZ Vaccine by DVI. Group C3 will undergo homologous CHMI with 3,200 PfSPZ Challenge (NF54), 3 weeks after vaccination.
  In case C3 shows <75% efficacy, verification phase will not be done.
  Interventions: Biological: PfSPZ Vaccine; Biological: PfSPZ Challenge (NF54)
- PfSPZ Challenge (7G8) dose finding - Group D1 (Experimental): n=3, one dose of 800 PfSPZ Challenge (7G8) by DVI.
  This is a dose finding study to assess safety, tolerability and infectivity of PfSPZ Challenge (7G8) administered DVI. CHMI with PfSPZ Challenge (7G8) will be done approximately at the same time as homologous CHMI to assess efficacy of immunization with PfSPZ Vaccine in the dose optimization phase. All volunteers receiving CHMI will be monitored by thick blood smear microscopy and qPCR until Day 28 or antimalarial treatment.
  Interventions: Biological: PfSPZ Challenge (7G8)
- PfSPZ Challenge (7G8) dose finding - Group D2 (Experimental): n=3, one dose of 1,600 PfSPZ Challenge (7G8) by DVI.
  This is a dose finding study to assess safety, tolerability and infectivity of PfSPZ Challenge (7G8) administered DVI. CHMI with PfSPZ Challenge (7G8) will be done approximately at the same time as homologous CHMI to assess efficacy of immunization with PfSPZ Vaccine in the dose optimization phase. All volunteers receiving CHMI will be monitored by thick blood smear microscopy and qPCR until Day 28 or antimalarial treatment.
  Interventions: Biological: PfSPZ Challenge (7G8)
- PfSPZ Challenge (7G8) dose finding - Group D3 (Experimental): n=3, one dose of 3,200 PfSPZ Challenge (7G8) by DVI.
  This is a dose finding study to assess safety, tolerability and infectivity of PfSPZ Challenge (7G8) administered DVI. CHMI with PfSPZ Challenge (7G8) will be done approximately at the same time as homologous CHMI to assess efficacy of immunization with PfSPZ Vaccine in the dose optimization phase. All volunteers receiving CHMI will be monitored by thick blood smear microscopy and qPCR until Day 28 or antimalarial treatment.
  Interventions: Biological: PfSPZ Challenge (7G8)
- Verification Phase - Group V1 (Experimental): n=12; optimal regimen from phase 1 - shortest, well tolerated safe schedule that provides >75% protection (5/6) against homologous CHMI (V1).
  Optimal & maximum regimens will be compared in this phase. The maximum regimen is a 3-dose regimen (Day 0, 7, 28) with highest well-tolerated PfSPZ Vaccine dose/injection (V2).
  Efficacy will be determined by repeat CHMI 3 and 8 weeks after last immunization. Inoculation of 2 CHMIs will be done about 35 days (5 weeks) apart.
  CHMI with PfSPZ Challenge (NF54) and CHMI with PfSPZ Challenge (7G8) will be administered in one of 2 sequences (NF54-7G8 or 7G8-NF54). Allocation to the 2 sequences will be double blind, random, at a 1:1 ratio and nested within the intervention groups (V1 and V2 PfSPZ Vaccine and placebo (P1 and P2)). CHMI will be done at a dose of 3,200 PfSPZ unless the dose escalation study of PfSPZ Challenge (7G8) indicates that a different dose would be preferable for 7G8.
  Interventions: Biological: PfSPZ Vaccine; Biological: PfSPZ Challenge (NF54); Biological: PfSPZ Challenge (7G8)
- Verification Phase - Group V2 (Experimental): n=12; maximum regimen from the phase 1 - 3-dose regimen (Day 0, 7 and 28) with highest well-tolerated PfSPZ Vaccine dose per injection (V2).
  Optimal & maximum regimens will be compared in this phase. The optimal regimen (shortest, well tolerated and safe schedule) that provides >75% protection (5/6) against homologous CHMI (V1).
  In case that shortest efficacious regimen during phase 1 is C3, 12 volunteers will be vaccinated and 6 volunteers will receive NS during this phase. In this case optimal regimen equals maximum regimen (3 x 2.7x10^6 PfSPZ). Group V2/P2 will not be immunized.
  Efficacy will be determined by repeat CHMI 3 and 8 weeks after last immunization. Inoculation of 2 CHMIs will be done about 35 days (5 weeks) apart.
  CHMI with PfSPZ Challenge (NF54) and CHMI with PfSPZ Challenge (7G8) will be administered as described in Group V1.
  Interventions: Biological: PfSPZ Vaccine; Biological: PfSPZ Challenge (NF54); Biological: PfSPZ Challenge (7G8)
- Verification Phase - Group P1 (Placebo Comparator): n=6; normal saline as placebo. This group will follow the regimen selected for Group V1.
  Efficacy of the vaccination regimen will be determined by CHMI which will be done by repeat CHMI three and eight weeks after the last immunization. Inoculation of the two CHMIs will be done approximately 35 days (5 weeks) apart.
  CHMI with PfSPZ Challenge (NF54) and CHMI with PfSPZ Challenge (7G8) will be administered as described in Group V1.
  Interventions: Biological: PfSPZ Challenge (NF54); Biological: PfSPZ Challenge (7G8); Other: Normal saline
- Verification Phase - Group P2 (Placebo Comparator): n=6; NS as placebo. This group will follow the regimen selected for Group V2.
  In case that shortest efficacious regimen during phase 1 is C3, 12 volunteers will be vaccinated and 6 volunteers will receive NS during this phase. In this case optimal regimen equals maximum regimen (3 x 2.7x10^6 PfSPZ). Group V2/P2 will not be immunized.
  Efficacy will be determined by repeat CHMI 3 and 8 weeks after the last immunization. Inoculation of the 2 CHMIs will be done about 35 days (5 weeks) apart.
  CHMI with PfSPZ Challenge (NF54) and CHMI with PfSPZ Challenge (7G8) will be administered as described in Group V1.
  Interventions: Biological: PfSPZ Challenge (NF54); Biological: PfSPZ Challenge (7G8); Other: Normal saline

INTERVENTIONS:
Biological: PfSPZ Vaccine — Aseptic, purified, vialed, cryopreserved, radiation-attenuated, Plasmodium falciparum sporozoites, strain NF54
  Arms: Optimization Phase - Group A; Optimization Phase - Group B1; Optimization Phase - Group B2; Optimization Phase - Group C1; Optimization Phase - Group C2; Optimization Phase - Group C3; Verification Phase - Group V1; Verification Phase - Group V2
Biological: PfSPZ Challenge (NF54) — Live, infectious, aseptic, purified, vialed, cryopreserved, Plasmodium falciparum sporozoites, strain NF54
  Arms: Optimization Phase - Group A; Optimization Phase - Group B1; Optimization Phase - Group B2; Optimization Phase - Group C1; Optimization Phase - Group C2; Optimization Phase - Group C3; Verification Phase - Group P1; Verification Phase - Group P2; Verification Phase - Group V1; Verification Phase - Group V2
Biological: PfSPZ Challenge (7G8) — Live, infectious, aseptic, purified, vialed, cryopreserved, Plasmodium falciparum sporozoites, strain 7G8
  Arms: PfSPZ Challenge (7G8) dose finding - Group D1; PfSPZ Challenge (7G8) dose finding - Group D2; PfSPZ Challenge (7G8) dose finding - Group D3; Verification Phase - Group P1; Verification Phase - Group P2; Verification Phase - Group V1; Verification Phase - Group V2
Other: Normal saline — 0.9% sodium chloride
  Arms: Verification Phase - Group P1; Verification Phase - Group P2

SUMMARY:
MAVACHE is a sequential dose and schedule optimization trial of intravenous immunization with PfSPZ Vaccine in 18 to 54 malaria-naïve, healthy adult volunteers receiving 9x10^5, 1.35x10^6, or 2.7x10^6 PfSPZ per dose and a total dose between 2.7x10^6 and 8.1x10^6 PfSPZ followed by CHMI with 3,200 fully infectious PfSPZ (PfSPZ Challenge).

PfSPZ Challenge (7G8) to assess vaccine efficacy, safety, tolerability and infectivity of ascending PfSPZ doses will be assessed in healthy, malaria-naïve volunteers.

DETAILED DESCRIPTION:
The study is to take place at Institut für Tropenmedizin, Eberhard Karls Universität Tübingen, Tübingen Germany.

The study has two phases: 1) dose optimization, and 2) regimen verification. In the first phase groups A, B1, B2, C1, C2 and C3 will be vaccinated sequentially in a pre-specified order, followed by homologous CHMI with 3,200 PfSPZ Challenge (NF54) three weeks after last vaccine injection.

Dose optimization phase A: 9x10^5 PfSPZ on Days 0, 7 and 28 (n = 6) B1: 1.35x10^6 PfSPZ on Days 0 and 7 (n = 6) B2: 1.35x10^6 PfSPZ on Days 0, 7, and 28 (n = 6) C1: 2.7x10^6 PfSPZ on Day 0 (n = 6) C2: 2.7x10^6 PfSPZ on Day 0 and 7 (n = 6) C3: 2.7x10^6 PfSPZ on Days 0, 7 and 28 (n = 6)

In parallel to CHMI with PfSPZ Challenge (NF54) during the optimization phase, a total of nine volunteers will receive either 800, 1,600 or 3,200 PfSPZ Challenge (7G8) (PfSPZ Challenge (7G8) dose finding) to assess safety, tolerability and infectivity of PfSPZ Challenge (7G8) in malaria-naïve healthy adult volunteers.

PfSPZ Challenge (7G8) dose finding/infection D1: 800 PfSPZ (n = 3) D2: 1,600 PfSPZ (n = 3) D3: 3,200 PfSPZ (n = 3)

Subsequently, the shortest efficacious regimen (V1) and a three-dose regimen (Day 0, 7 and 28) of the highest safe dose (V2) will be selected and verified against placebo (normal saline (NS)). Groups V1 and V2 will be vaccinated at approximately the same time and undergo repeat CHMI three and eight weeks after the last immunization. Volunteers will either receive PfSPZ Vaccine or NS as placebo. Allocation will be random and double blind. Repeat CHMI will be done with PfSPZ Challenge (NF54) and PfSPZ Challenge (7G8), given in a randomized sequence. All immunizations are given by direct venous inoculation (DVI).

Regimen verification phase V1: Shortest efficacious regimen (n = 12) against placebo (n = 6) V2: Maximum regimen (n = 12) against placebo (n = 6) P1: Placebo for V1 group (n=6) P2 Placebo for V2 group (n=6)

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 to 45 years
* Able and willing (in the Investigator's opinion) to comply with all study requirements
* Willing to allow the investigators to discuss the volunteer's medical history with their general practitioner ('Hausarzt' in German) if required
* Residence in Tübingen or surroundings for the period of the trial
* Women only: Must agree to practice continuous effective contraception for the duration of the study (a method which results in a failure rate less than 1% per year)
* Agreement to refrain from blood donation during the course of the study and after the end of their involvement in the study according to the local and national blood banking eligibility criteria (currently there is a four year restriction in Germany)
* Written informed consent to receive PfSPZ products:
* Optimization phase: PfSPZ Vaccine for immunization and PfSPZ Challenge (NF54) for CHMI
* PfSPZ Challenge (7G8) dose finding: PfSPZ Challenge (7G8) for CHMI
* Verification phase: PfSPZ Vaccine for immunization, PfSPZ Challenge (NF54) and PfSPZ Challenge (7G8) for CHMI
* Reachable (24/7) by mobile phone during the immunization and CHMI period
* Willingness to take a curative antimalarial regimen following CHMI
* Agreement to stay overnight for observation during the period of intensive follow-up post-challenge if required
* Answer all questions on the informed consent quiz correctly
* A body mass index <35

Exclusion Criteria:

* History of P. falciparum malaria
* Planned travel to malaria endemic areas before end of CHMI (28 days after CHMI)
* Use of systemic antibiotics with known antimalarial activity within 30 days of study enrollment (e.g. trimethoprim-sulfamethoxazole, doxycycline, tetracycline, clindamycin, erythromycin, fluoroquinolones, or azithromycin)
* Receipt of an investigational product in the 30 days preceding enrollment, or planned receipt during the study period
* Prior receipt of a malaria vaccine
* Immunization with more than three other vaccines within the past four weeks
* HIV infection
* Any confirmed or suspected immunosuppressive or immunodeficient state, asplenia, recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed)
* Use of immunoglobulins or blood products within 3 months prior to enrolment
* Known or suspected hemolytic disease or presence of hemoglobinopathies
* Pregnancy, lactation or intention to become pregnant during the study
* Contraindications to the use of the following antimalarial medications: atovaquoneproguanil, artemether-lumefantrine or mefloquine
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ)
* History of serious psychiatric condition that may affect participation in the study (including but not restricted to organic, including symptomatic, mental disorders [ICD-10 code: F00-F09], schizophrenia, schizotypal and delusional disorders [F20-F29], mood (affective) disorders [F30-F39], mental retardation [F70-F79], Disorders of psychological development [F80-F89] or any other psychiatric condition that required hospitalization or psychiatric treatment over an extended period).
* Any other serious chronic illness requiring hospital specialist supervision
* Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 60 g (men) or 40 g (women) per day or a carbohydrate deficient transferrin (CDT) level ≥2.5%
* Suspected or known injecting drug abuse in the 5 years preceding enrollment
* Positive for hepatitis B surface antigen (HBs-antigen)
* Seropositive for hepatitis C virus (antibodies to HCV)
* Falling in moderate risk or higher categories for fatal or non-fatal cardiovascular event within 5 years (>10%) determined by non-invasive criteria for cardiac risk
* Abnormal electrocardiogram on screening: pathologic Q wave and significant ST-T wave changes, left ventricular hypertrophy, clinically significant arrhythmias, left bundle branch block, secondary or tertiary A-V heart block
* A QT/QTcB interval >450 ms
* Volunteers unable to be closely followed for social, geographic or psychological reasons
* Any clinically significant abnormal finding on biochemistry or hematology blood tests, urine analysis or clinical examination
* History of seizure (except isolated and uncomplicated febrile convulsion at childhood)
* Any other significant disease, disorder or finding which, in the opinion of the investigator, may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2016-08-29 (Actual); Primary Completion 2018-10-19 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Number or occurrence of at least possibly related Grade 3 AEs and serious adverse events (SAEs) for PfSPZ Vaccine | Around 14 months (from day of first immunization through study completion)
  Number or occurrence of at least possibly related Grade 3 AEs and SAEs from time of first administration of PfSPZ Vaccine to the end of the follow-up period.
PfSPZ Challenge (7G8) dose finding - Number or occurrence of at least possibly related Grade 3 AEs and SAEs | Around 140 days (from day of first PfSPZ Challenge (7G8) CHMI through end of follow-up)
  Number or occurrence of at least possibly related Grade 3 AEs and SAEs from time of first administration of PfSPZ Challenge (7G8) to the end of the follow-up period.

SECONDARY OUTCOMES:
Number of adverse events following immunization (AEFI) for PfSPZ Vaccine | About 7 weeks (from day of first vaccination until 3 weeks after last vaccination)
  Number of adverse events following immunization (AEFI) from time of first administration of PfSPZ Vaccine to first administration of PfSPZ Challenge for CHMI consistent with a causal relationship.
Proportion of volunteers who become parasitemic will be recorded, detected by thick blood film microscopy or qPCR | Up to 4 weeks (from day of CHMI until 28 days)
  Thick blood film microscopy and quantitative polymerase chain reaction (qPCR) assays will be performed during CHMI follow-up. The proportion of volunteers who become parasitemic will be recorded, detected by thick blood film microscopy or qPCR, within 28 days following CHMI with 3,200 PfSPZ, given either as a single dose of 3,200 PfSPZ Challenge (NF54) (optimization phase) or as two subsequent injections of 3,200 PfSPZ Challenge (NF54) and PfSPZ Challenge (7G8), respectively in the verification phase.
Proportion of volunteers who do not become parasitemic (protected) against homologous (NF54) and heterologous (7G8) CHMI, respectively. | About 28 days (from day of first CHMI till 28 days)
  This endpoint can only be assessed during the verification phase of the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Mordmüller, MD, Principal Investigator — Institute of Tropical Medicine, University of Tuebingen, Wilhelmstr. 27, Germany
Locations (1):
- Institute of Tropical Medicine, University of Tuebingen, Wilhelmstr. 27, Tübingen, Germany

REFERENCES:
- [Derived] Wichers-Misterek JS, Krumkamp R, Held J, von Thien H, Wittmann I, Hoppner YD, Ruge JM, Moser K, Dara A, Strauss J, Esen M, Fendel R, Sulyok Z, Jeninga MD, Kremsner PG, Sim BKL, Hoffman SL, Duffy MF, Otto TD, Gilberger TW, Silva JC, Mordmuller B, Petter M, Bachmann A. The exception that proves the rule: Virulence gene expression at the onset of Plasmodium falciparum blood stage infections. PLoS Pathog. 2023 Jun 29;19(6):e1011468. doi: 10.1371/journal.ppat.1011468. eCollection 2023 Jun. PMID 37384799
- [Derived] Mordmuller B, Sulyok Z, Sulyok M, Molnar Z, Lalremruata A, Calle CL, Bayon PG, Esen M, Gmeiner M, Held J, Heimann HL, Woldearegai TG, Ibanez J, Flugge J, Fendel R, Kreidenweiss A, Kc N, Murshedkar T, Chakravarty S, Riyahi P, Billingsley PF, Church LWP, Richie TL, Sim BKL, Hoffman SL, Kremsner PG. A PfSPZ vaccine immunization regimen equally protective against homologous and heterologous controlled human malaria infection. NPJ Vaccines. 2022 Aug 23;7(1):100. doi: 10.1038/s41541-022-00510-z. PMID 35999221